CLINICAL TRIAL: NCT05293483
Title: The Impact of Hospital Care for COVID-19 on the Prevalence of Multidrug-resistant Microorganisms Among Patients Compared to Non-COVID-19 Hospital Care in Limited-resource Hospitals in Indonesia
Brief Title: The Impact of Covid-19 Hospital Care on the Prevalence of MDRO in Indonesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: British Society for Antimicrobial Chemotherapy (Other); University of Brawijaya (Other); Saiful Anwar Hospital (Other); Ngudi Waluyo Hospital (Unknown)
Responsible Party: Principal Investigator, Juliëtte Severin, Associate professor, Medical coordinator Unit infection prevention, Erasmus Medical Center
Other Study IDs: 400/213/K.3/302/2021
Record Dates: First submitted 2022-03-22; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Antibiotic Resistant Infection; COVID-19
Keywords: Antimicrobial resistant; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — The bacterial DNA will be extracted from multidrug resistant bacteria isolates obtained from sputum, blood, pus, and urine of patients hospitalized in both COVID-19 wards and non-COVID-19 wards.

GROUPS / COHORTS (2):
- COVID-19
- non-COVID-19

SUMMARY:
The effect of the COVID-19 pandemic on the emergence and spread of antibiotic-resistant bacteria is largely unknown, especially in low-resource settings. We aim to investigate the prevalence and relatedness of multidrug-resistant bacteria among patients in both COVID-19 and non-COVID-19 wards in two hospitals in Indonesia. Bacterial isolates will be collected from clinical sample and by screening of patients at discharge followed by 30 days after discharge. Aspects of hospital care that may be different in COVID-19 wards versus non-COVID-19 wards and that are considered important determinants for antimicrobial resistance (AMR) will be measured: hand hygiene compliance, use of personal protective equipment, and antibiotic use. Comparison of these data from COVID-19 wards to non-COVID-19 wards will increase our understanding of multidrug-resistant bacteria and provide further insight into the effect of interventions for AMR.

The hypothesis of this study are: 1) the prevalence of multidrug-resistant bacteria in COVID-19 wards is higher than non-COVID-19 wards; 2) there is a relatedness of multidrug-resistant bacteria circulating either in the COVID-19 wards or non-COVID-19 wards; 3) the hand-hygiene compliance is lower in the COVID-19 wards than non-COVID-19 wards, however the personal protective equipment use compliance is higher in the COVID-19 wards than non-COVID-19 wards; 4) the antibiotic use in non-COVID-19 wards is better qualitatively; 5) the use of Ciprofloxacin, Gentamicin, and Ceftriaxone in non-COVID-19 wards is higher than in COVID-19 wards.

DETAILED DESCRIPTION:
The overall objective of the study is to reveal the impact of hospital care for COVID-19 patients on the prevalence of MDRO among COVID-19 patients, compared to non-COVID-19 hospital care and the prevalence of MDRO among non-COVID-19 patients, with its underlying determinants in limited-resource hospitals in Indonesia.

Specific aims of the study:

1. To measure the prevalence of MDRO in the COVID-19 wards compared to non-COVID-19 wards.
2. To investigate the transmission of the most prevalent MDRO in the COVID-19 wards compared to non-COVID-19 wards.
3. To analyze the hand hygiene compliance and use of PPE in COVID-19 wards compared to non-COVID-19 wards.
4. To analyze the antibiotic use in COVID-19 wards compared to non-COVID-19 wards.

Design of the study:

A prospective, observational cohort study will be performed in both COVID-19 wards and non-COVID-19 wards of a secondary care and a tertiary care hospital in the province of East Java in Indonesia. Both intensive care units (ICUs) and non-ICUs will be used. The tertiary care hospital in Malang is the Dr. Saiful Anwar hospital with 882 beds. Currently, 80 COVID-19 patients are admitted each month. The secondary care hospital has 250 beds, and approximately 25 COVID-19 patients are admitted each month.

The specific aims will be addressed as follows:

1. MDRO prevalence

   The following MDROs will be included: MRSA, ESBL-producing Escherichia coli, ESBL-producing and carbapenemase-producing K. pneumoniae, carbapenem-resistant P. aeruginosa, and carbapenem-resistant A. baumannii. These will be searched for and collected via two approaches:
   1. Detection by routine clinical cultures from patients during their hospital stay, both in the COVID-19 wards and non-COVID-19 wards. Blood, lower respiratory tract specimens, pus, and urine will be eligible for inclusion in the study. Identification and antibiotic susceptibility testing of the MDROs will be performed by the Vitek2 system. Demographic data and data on medical history, in-hospital mortality, length of stay, and antibiotic use will be collected from the medical records, according to the national regulations of medical research. The overall number of clinical cultures and their results will be collected for prevalence calculations (WHOnet).
   2. As results from clinical cultures only reveal the tip of the MDRO iceberg, adult patients will be actively screened for MDRO carriage on the day of discharge and 30 days post-discharge from the COVID-19 ward and the non-COVID-19 ward, after informed consent. Discharge screening has been used as an approach in previous studies, and shown to be useful to detect MDRO transmission in the hospital. Screening on admission would be useful as well, but is not feasible on the COVID-wards due to workload when a patient is ill and needs immediate care. The 30-day post-discharge screening is a novel approach which may reveal MDROs that are still undetectable (i.e. in lowloads) in or on the patient's body on the moment of discharge, for example due to antibiotic use. All adult patients discharged from these wards are eligible for inclusion in the study. However, patients discharged within 48 hours of admission and patients who either live outside the city of Malang or their address is unclear are excluded. The 30-day post-discharge screening can be organized via the local public health centre.

   Sample size consideration:

   We expect to include at least 500 COVID-19 patients and 500 non-COVID-19 patients for MDRO detection from clinical culture, and at least 120 COVID-19 and 120 non-COVID-19 patients for active screening.

   Microbiological methods:

   Anterior nares and rectal swabs will be taken from each patient for discharge and post-discharge screening using sterile cotton swabs and transported to the laboratory in Amies transport medium for further processing within 24 hours of sampling. Isolation and identification of MDROs from the swabs will be performed as previously described. Confirmation of ESBL production will be done with the combination disk test, carbapenemase production with the CIM test. Isolates will be stored in duplicate as was done in our previous studies.
2. Analysis of MDRO transmission Detection of common resistance genes (i.e. mecA, blaNDM etc.) will be conducted by polymerase chain reaction. The clonality of MDROs will be evaluated for the most prevalent MDROs: by spa/MLVA typing (MRSA) and whole genome sequencing (Gram-negative MDRO; Illumina/nanopore).
3. Hand hygiene and PPE The direct observation method will be applied to establish hand hygiene compliance rate and use of PPE (gloves, gowns, masks). This will be done monthly during the one year period that bacterial isolates are collected.
4. Antibiotic use analysis Qualitative evaluation of antibiotic use will be performed by the Gyssens' algorithm and subsequent comparison of COVID-19 patients and non-COVID-19 patients either with or without MDRO infection or colonization. Furthermore, the DDD value of ceftriaxone, gentamicin, and ciprofloxacin will be compared.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients discharged from Covid wards and non Covid wards (ICU and internal medicine wards)

Exclusion Criteria:

* Patients discharged within 48 hours of admission
* Patients who either live outside the city of Malang or their address is unclear

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients will be actively screened for MDRO carriage on the day of discharge and 30 days post-discharge from the COVID-19 ward and the non-COVID-19 ward (ICU and internal medicine wards)
Sampling Method: Probability Sample
Enrollment: 1110 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-12-07 (Estimated); Study Completion 2023-03-07 (Estimated)

PRIMARY OUTCOMES:
Multidrug resistant bacteria prevalence | One year
  MRSA, ESBL-producing Escherichia coli, ESBL-producing and carbapenemase-producing K. pneumoniae, carbapenem-resistant P. aeruginosa, and carbapenem-resistant A. baumannii will be searched for via two approaches including clinical culture and active screening among COVID-19 patients and non -COVID-19 patients.
Multidrug resistant bacteria transmission | One year
  Detection of common resistance genes (i.e. mecA, blaNDM etc.) will be conducted by polymerase chain reaction. The clonality of MDROs will be evaluated for the most prevalent MDROs: by spa/MLVA typing (MRSA) and whole genome sequencing (Gram-negative MDRO; Illumina/nanopore).
Hand Hygiene and Personal Protective Equipment Use Compliance | One year
  The direct observation method will be applied to establish hand hygiene compliance rate and use of PPE (gloves, gowns, masks).
Antibiotic use analysis | One year
  Qualitative evaluation of antibiotic use will be performed by the Gyssens' algorithm and subsequent comparison of COVID-19 patients and non-COVID-19 patients either with or without MDRO infection or colonization. Furthermore, the DDD value of ceftriaxone, gentamicin, and ciprofloxacin will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Dewi Santosaningsih, PhD, Principal Investigator — Dpt Clin Microbiology, Faculty of Medicine, Brawijaya University/Dr Saiful Anwar Hospital, Malang, Indonesia
Locations (2):
- Indonesia (2):
  - Ngudi Waluyo hospital, Blitar, East Java
  - dr. Saiful Anwar hospital, Malang, East Java

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saharman YR, Karuniawati A, Sedono R, Aditianingsih D, Sudarmono P, Goessens WHF, Klaassen CHW, Verbrugh HA, Severin JA. Endemic carbapenem-nonsusceptible Acinetobacter baumannii-calcoaceticus complex in intensive care units of the national referral hospital in Jakarta, Indonesia. Antimicrob Resist Infect Control. 2018 Jan 12;7:5. doi: 10.1186/s13756-017-0296-7. eCollection 2018. PMID 29344351
- [Background] Hsu LY, Apisarnthanarak A, Khan E, Suwantarat N, Ghafur A, Tambyah PA. Carbapenem-Resistant Acinetobacter baumannii and Enterobacteriaceae in South and Southeast Asia. Clin Microbiol Rev. 2017 Jan;30(1):1-22. doi: 10.1128/CMR.masthead.30-1. Epub 2016 Oct 19. PMID 27795305
- [Background] Clancy CJ, Nguyen MH. Coronavirus Disease 2019, Superinfections, and Antimicrobial Development: What Can We Expect? Clin Infect Dis. 2020 Dec 17;71(10):2736-2743. doi: 10.1093/cid/ciaa524. PMID 32361747
- [Background] Rawson TM, Moore LSP, Zhu N, Ranganathan N, Skolimowska K, Gilchrist M, Satta G, Cooke G, Holmes A. Bacterial and Fungal Coinfection in Individuals With Coronavirus: A Rapid Review To Support COVID-19 Antimicrobial Prescribing. Clin Infect Dis. 2020 Dec 3;71(9):2459-2468. doi: 10.1093/cid/ciaa530. PMID 32358954
- [Background] Lestari ES, Severin JA, Filius PM, Kuntaman K, Duerink DO, Hadi U, Wahjono H, Verbrugh HA; Antimicrobial Resistance in Indonesia: Prevalence and Prevention (AMRIN). Antimicrobial resistance among commensal isolates of Escherichia coli and Staphylococcus aureus in the Indonesian population inside and outside hospitals. Eur J Clin Microbiol Infect Dis. 2008 Jan;27(1):45-51. doi: 10.1007/s10096-007-0396-z. Epub 2007 Oct 13. PMID 17934766
- [Background] Santosaningsih D, Santoso S, Budayanti NS, Kuntaman K, Lestari ES, Farida H, Hapsari R, Hadi P, Winarto W, Milheirico C, Maquelin K, Willemse-Erix D, van Belkum A, Severin JA, Verbrugh HA. Epidemiology of Staphylococcus aureus harboring the mecA or Panton-Valentine leukocidin genes in hospitals in Java and Bali, Indonesia. Am J Trop Med Hyg. 2014 Apr;90(4):728-34. doi: 10.4269/ajtmh.13-0734. Epub 2014 Feb 24. PMID 24567320
- [Background] Saharman YR, Pelegrin AC, Karuniawati A, Sedono R, Aditianingsih D, Goessens WHF, Klaassen CHW, van Belkum A, Mirande C, Verbrugh HA, Severin JA. Epidemiology and characterisation of carbapenem-non-susceptible Pseudomonas aeruginosa in a large intensive care unit in Jakarta, Indonesia. Int J Antimicrob Agents. 2019 Nov;54(5):655-660. doi: 10.1016/j.ijantimicag.2019.08.003. Epub 2019 Aug 7. PMID 31398483
- [Background] Saharman YR, Karuniawati A, Sedono R, Aditianingsih D, Goessens WHF, Klaassen CHW, Verbrugh HA, Severin JA. Clinical impact of endemic NDM-producing Klebsiella pneumoniae in intensive care units of the national referral hospital in Jakarta, Indonesia. Antimicrob Resist Infect Control. 2020 May 11;9(1):61. doi: 10.1186/s13756-020-00716-7. PMID 32393386
- [Background] van der Zwaluw K, de Haan A, Pluister GN, Bootsma HJ, de Neeling AJ, Schouls LM. The carbapenem inactivation method (CIM), a simple and low-cost alternative for the Carba NP test to assess phenotypic carbapenemase activity in gram-negative rods. PLoS One. 2015 Mar 23;10(3):e0123690. doi: 10.1371/journal.pone.0123690. eCollection 2015. PMID 25798828
- [Background] Santosaningsih D, Erikawati D, Santoso S, Noorhamdani N, Ratridewi I, Candradikusuma D, Chozin IN, Huwae TECJ, van der Donk G, van Boven E, Voor In 't Holt AF, Verbrugh HA, Severin JA. Intervening with healthcare workers' hand hygiene compliance, knowledge, and perception in a limited-resource hospital in Indonesia: a randomized controlled trial study. Antimicrob Resist Infect Control. 2017 Feb 16;6:23. doi: 10.1186/s13756-017-0179-y. eCollection 2017. PMID 28239452